CLINICAL TRIAL: NCT05615675
Title: Immersive Audiovisual Distraction With Virtual Reality (VR) in Prone Procedures in the Interventional Pain Clinic
Brief Title: Virtual Reality (VR) for Prone Pain Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1919687
Record Dates: First submitted 2022-09-26; First posted 2022-11-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Patients undergo prone pain procedure with virtual reality distraction
  Interventions: Other: Virtual Reality Headset
- Control (No Intervention): Patients undergo prone pain procedure without virtual reality distraction

INTERVENTIONS:
Other: Virtual Reality Headset — Patient uses a virtual reality headset and support during prone pain procedure
  Other Names: Oculus Quest Virtual Reality Headset
  Arms: Virtual Reality

SUMMARY:
The purpose of this study is to evaluate the effectiveness of virtual reality (VR) distraction in patients undergoing interventional pain procedures in the prone position. VR has been shown to improve patient experience during interventional pain procedures, however, many of these procedures are done in the prone position making VR a challenge. This study will evaluate the effect of a VR headset and support in patients undergoing prone interventional pain procedures compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or older, who are referred to University of California Davis Pain Medicine Clinic and require an interventional pain procedure
* English speaking and with the ability to understand oral and written instructions

Exclusion Criteria:

* Pregnant women
* Prisoners
* Patients who have high risk of motion sickness, seizure disorder, or visual/hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Anxiety Score | Immediately before procedure
  State-Trait Anxiety Inventory (Self-reported anxiety instrument containing two separate 2-item subscales that measure trait (baseline) and state (situational) anxiety; Total range 20 to 80 with higher scores indicating greater anxiety).
Anxiety Score | Immediately after procedure
  State-Trait Anxiety Inventory (Self-reported anxiety instrument containing two separate 2-item subscales that measure trait (baseline) and state (situational) anxiety; Total range 20 to 80 with higher scores indicating greater anxiety).

SECONDARY OUTCOMES:
Anxiety Score | Immediately before procedure, during procedure, and immediately after procedure
  Anxiety score on an 11-point numerical rating scale (Total range 0-10 with higher scores indicating greater pain)
Pain Score | Immediately before procedure, during procedure, and immediately after procedure
  Pain score on an 11-point numerical rating scale (Total range 0-10 with higher scores indicating greater pain)
Global Impression of Change | Immediately after procedure
  Global Impression of Change on a 7-point scale (Lower scores indicating decline in clinical status, and higher scores indicating improvement in clinical status)
Patient Experience Satisfaction | Immediately after procedure
  Experience Satisfaction on an 11-point scale (Total range 0-10 with higher scores indicating higher patient experience satisfaction)
Sedation Requirements | During course of procedure
  Amount of benzodiazepines and opioid medications given

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jung, MD MBA, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Interventional Pain Clinic, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No